CLINICAL TRIAL: NCT02050191
Title: The Primary Goal of the Phase I Research Was to Demonstrate Feasibility of Creating and Running an Incentive-based Wellness Portal for a Local Community (Princeton, NJ) That Involved Designing the System, Building a Prototype, Testing the System, and Assessing User Acceptance.
Brief Title: Community Web Health Portal for Diabetes Prevention
Acronym: NnoLEDGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Griffin Hospital (Other)
Collaborators: Viocare, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2005-10
Record Dates: First submitted 2012-10-10; First posted 2014-01-30 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Obesity; Health Knowledge
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- program feasibility (No Intervention)
  Interventions: Behavioral: www.princetonlivingwell.com

INTERVENTIONS:
Behavioral: www.princetonlivingwell.com

SUMMARY:
This study supports the development of a diabetes prevention and control community web portal. The portal will feature an innovative personalized impediment profiling tool and reward program. The program, "Nutrition Navigation on-Line Edge," or NnoLEDGE, will be used by community consortiums for weight loss and diabetic health interventions within their communities.

The Specific Aims are:

1. Recruitment of local community organizations to participate as a community health consortium
2. Development of a comprehensive community health web portal consisting of a web portal, impediment profiler, community toolbox, and rewards system
3. Final evaluation of the system with regard to participants' attitudes and perceptions of using NnoLEDGE as a tool for weight control and diabetes prevention to determine feasibility.

ELIGIBILITY:
Inclusion Criteria:

* can read and write English

Exclusion Criteria:

* cannot read and write Engish

Ages: 18 Years to 70 Years | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-07; Primary Completion 2009-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
attitudes and perceptions re: feasibility of web portal | 2 months
  Subjects will complete surveys aimed at assessing their attitudes and perceptions of the feasibility of the use of the nNoledge tool for weight control and prevention of diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Rick Weiss, MS, Principal Investigator — Viocare, Inc.